CLINICAL TRIAL: NCT06126263
Title: Comparative Effectiveness of Adjunctive Clindamycin Versus Linezolid for β-lactam Treated Patients With Invasive Group A Streptococcal Infections: A Target Trial Emulation
Brief Title: Adjunctive Clindamycin Versus Linezolid for β-lactam Treated Patients With Invasive Group A Streptococcal Infections
Acronym: iGASAntitox
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Sameer Kadri, M.D., Tenure Track Investigator, National Institutes of Health Clinical Center (CC)
Other Study IDs: BD022389
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Streptococcal Sepsis; Invasive Group A Beta-Haemolytic Streptococcal Disease; Necrotizing Soft Tissue Infection; Infection, Bloodstream; Infection, Bacterial; Streptococcal Toxic Shock Syndrome
Keywords: Invasive GAS; necrotizing soft tissue infection; streptococcal toxic shock syndrome; linezolid; clindamycin; anti-toxin therapy
MeSH Terms: conditions — Sepsis; Bacterial Infections | interventions — Linezolid; Clindamycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Linezolid — Adjunctive antitoxin therapy
Drug: Clindamycin — Adjunctive antitoxin therapy

SUMMARY:
This study aims to emulate a hypothetical target pragmatic multi-center, non-blinded trial of adult inpatients in the PINC AITM dataset with B-lactam treated culture confirmed monomicrobial invasive Group A streptococcus (GAS) between the years 2015-2021

ELIGIBILITY:
Inclusion Criteria:

* Adult inpatients patients (=> 18 y of age)
* Monomicrobial Group A streptococcus invasive infection
* Primary therapy with a B-lactam agent (initiated before or on same day as adjunctive anti-toxin therapy)

Exclusion Criteria:

* Patients with a polymicrobial GAS culture (non-GAS organisms identified on eligibility GAS culture)
* Patients who received linezolid but have a documented linezolid resistant isolate
* Patients with GAS infections of non-sterile non-invasive sites (i.e sites which do not meet above mentioned inclusion criteria) which include but not limited to the lower urinary tract, upper respiratory tract
* Patient with concomitant MSSA/MRSA invasive infection (+/- seven days of index GAS eligibility culture)
* Patients who receive both anti-toxin agents (violation of protocol)
* Patient who do not complete at least 3 days of B-lactam (violation of protocol)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult inpatients with culture confirmed proven or probable invasive monomicrobial GAS in the PINC AI (TM) Database admitted between 2015-2021 who receive a β-lactam therapy for a minimum of 3 days within 3 days of culture will be eligible for inclusion in the emulated trial. Patient will be included if they then receive an anti-toxin therapy within 3 days of culture being drawn, as long as B-lactam therapy has been initiated prior or on the same day as antitoxin therapy.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
In hospital mortality or discharge to hospice | Hospital stay
  In hospital mortality or discharge to hospice

SECONDARY OUTCOMES:
Length of stay among survivors | Hospital stay
  Duration of hospitalization among surviving participants
Clostridioides difficile infection | Within hospital stay of interest
  C. difficile positive (PCR or antigen) result within same encounter downstream of the antitoxin therapy within 30 days and/or presence of a non present on admission (POA) C. difficile diagnosis code in conjugation with receipt of C. difficile therapy (PO/rectal vancomycin or PO fidaxomicin or IV metronidazole)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Babiker, Principal Investigator — Emory University
Locations (1):
- National Institutes of Health Clinical Center (primary center conducting large database study), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/63/NCT06126263/Prot_SAP_000.pdf